CLINICAL TRIAL: NCT00420888
Title: A Randomized, Open-label, Multi-center, Phase II/III Study on Treatment With ABR-217620/Naptumomab Estafenatox Combined With IFN-alpha vs. IFN-alpha Alone in Patients With Advanced Renal Cell Carcinoma.
Brief Title: ABR-217620/Naptumomab Estafenatox With Interferon-alpha (IFN-alpha) Compared to IFN-alpha Alone in Patients With Advanced Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Active Biotech AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06762004
Record Dates: First submitted 2007-01-09; First posted 2007-01-11 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2014-06

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — naptumomab estafenatox; Interferon-alpha

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Safety group (Experimental): 6-12 patients
  Interventions: Drug: ABR-217620/naptumomab estafenatox; Drug: IFN-alpha
- 1 (Experimental)
  Interventions: Drug: ABR-217620/naptumomab estafenatox; Drug: IFN-alpha
- 2 (Other): Standard treatment with IFN-alpha without add-on of ABR-217620/naptumomab estafenatox
  Interventions: Drug: IFN-alpha

INTERVENTIONS:
Drug: ABR-217620/naptumomab estafenatox — 10 mcg/kg or 15 mcg/kg, 5 minute bolus intravenous injection on 4 consecutive days / 8 week cycle repeated 3 times
  Other Names: naptumomab estafenatox
  Arms: 1; Safety group
Drug: IFN-alpha — 3 MIU, 6 MIU, and 9 MIU, subcutaneous or intramuscular injection 3 times / week
  Other Names: Referon-A

SUMMARY:
The drug ABR-217620/naptumomab estafenatox is a fusion of two proteins, one that recognizes tumor cells and one that triggers an attack on the tumor cells by activating some white blood cells belonging to the body's normal immune system. This results in an accumulation of white blood cells in the cancer that can fight the cancer. This study will compare the safety and effectiveness (assessed by tumor status and survival) of ABR-217620/naptumomab estafenatox when given with standard therapy IFN-alpha to IFN-alpha alone in patients with advanced renal cell carcinoma (RCC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed RCC (clear cell and papillary types)
* Metastatic or inoperable locally advanced RCC
* Eligible for therapy with IFN-alpha.
* Measurable disease defined by at least 1 measurable lesion on CT scan (lesion diameter greater than or equal to 2.0 cm by a standard CT scanner or greater than or equal to 1.0 cm by a spiral CT scanner)
* Favorable or moderate risk group prognosis by MSKCC (Motzer) criteria (score 0-2)
* Karnofsky performance status greater than or equal to 70
* Age greater than or equal to 18
* Life expectancy greater than 3 months
* Baseline blood counts:

  * Absolute neutrophil count (ANC) greater than or equal to 1.5 x 10^9/L
  * Platelets greater than or equal to 100 x 10^9/L
  * Haemoglobin greater than or equal to 100 g/L
* Baseline blood chemistry levels:

  * Creatinine less than or equal to 1.5 x upper limit of normal (ULN)
  * Bilirubin less than or equal to 2 x ULN
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than or equal to 2.5 x ULN. AST and ALT allowed less than or equal to 5 x ULN for patients with liver metastases.
* If fertile, patient will use effective method of contraception throughout the study
* Willing and able to comply with the treatment and follow-up visits and examinations
* Capable of understanding the parameters in the protocol and able to sign a written consent form

Exclusion Criteria:

* Pregnant or breastfeeding women
* Serious uncontrolled medical disorder or active infection ongoing or resolved within 2 weeks before first dose of study drug and that the investigator believes would impair the patient's ability to receive study drug
* History of malignancy within 5 years or concurrent malignancy, except successfully treated non-melanoma skin cancer, cervical cancer in situ, ductal carcinoma in situ or lobular carcinoma in situ of breast may be included
* History and/or signs of parenchymal brain metastases
* Significant cardiac disease including: history (within 6 months) or current unstable angina pectoris, congestive heart failure (NYHA stage III-IV), myocardial infarction within 12 months, or uncontrolled arterial hypertension.
* History of stroke within 5 years and/or transient ischemic attack within 6 months.
* Acute illness or evidence of infection, including unexplained fever (>100.5ºF or 38.1ºC) within 2 weeks before start of treatment
* Treatment with biological response modifiers within 3 weeks prior to the start of treatment and up to the End-of-Study visit
* Treatment with beta-blockers, including topical therapy for glaucoma, within 5 days before start of treatment and during the 4-day ABR-217620/naptumomab estafenatox treatment
* Treatment with systemic corticosteroids within 2 weeks before start of treatment or likely need for such treatment during the study
* Active autoimmune disease requiring therapy or any history of systemic lupus erythematosus or rheumatoid arthritis
* Known positive serology for HIV
* Chronic hepatitis with advanced, decompensated hepatic disease or cirrhosis of the liver or history of chronic virus hepatitis or known virus carrying; patients who recovered from Hepatitis A are allowed
* Treatment with anticoagulants within 2 weeks before start of treatment, except when used to maintain the patency of a central or peripheral venous line
* Radiotherapy less than 4 weeks before start of treatment
* Major surgery or tumor embolization less than 4 weeks before start of treatment
* Previous exposure to murine monoclonal antibodies or known hypersensitivity to murine proteins
* Currently on renal dialysis treatment
* Known allergy or hypersensitivity to aminoglycosides and kanamycin
* Previous systemic anti-tumor therapy for RCC (including immunotherapy with IFN-alpha or IL-2 or any chemotherapy) except sunitinib or other oral antiangiogenic therapy
* Participation in any study with investigational drugs for RCC within 6 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 526 (Actual)
Dates: Start 2007-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Time to death | every 12 weeks, including after a maximum of 18 months of study treatment

SECONDARY OUTCOMES:
Progression-free survival time | every 12 weeks for the 18-month treatment period and also every 12 weeks after the treatment period
Objective tumor response rate | every 12 weeks for the 18-month treatment period
Best overall response | every 12 weeks for the 18-month treatment period
Duration of response | every 12 weeks for the 18-month treatment period
Changes in sum of target lesions | every 12 weeks for the 18-month treatment period
Immunological response in patients on combined treatment of ABR-217620/naptumomab estafenatox and IFN-alpha | Weeks 1, 9, 17, 25, 73
Vital signs | every visit through Week 25, plus Week 73
Physical measurements | Weeks 1, 9, 17, 25, 73
Adverse events | every visit through Week 73
Laboratory safety assessments | Weeks 1, 2, 3, 5, 9, 10, 13, 17, 18, 21, 25, and 73
Pharmacokinetic parameters of ABR-217620/naptumomab estafenatox | Weeks 1, 9, and 17

CONTACTS AND LOCATIONS:
Overall Officials: Thore Nederman, PhD, Study Director — Active Biotech AB
Locations (51):
- Bulgaria (6):
  - Department of Chemotherapy, University General Hospital for Active Treatment "Georgi Stranski", Pleven
  - 1st Internal Department District Dispensary for Cancer Diseases with Inpatient Hospital, Plovdiv
  - Multifile Hospital "Aleksandrovska", Urology Clinic, Department of Oncourology, Sofia
  - Oncology Clinic, University General Hospital for Active Treatment "Tzaritza Yoanna", Sofia
  - Urology Clinic, General Hospital for Active Treatment "St. Anna", Varna
  - Department of Chemotherapy, Inter-district Dispensary for Cancer Diseases with Inpatient Hospital, Veliko Tarnovo
- Romania (8):
  - Fundeni Clinical Institute - Urology Department, Bucharest
  - Dinu Uromedica, Bucharest
  - "Prof. Dr. Th. Burghele" Clinical Hospital, Urology Clinic, Bucharest
  - "I. Chiricuta" Institute of Oncology, Cluj-Napoca
  - E-URO Medical Center, Cluj-Napoca
  - Provita Center SRL, Constanța
  - Sibiu Clinical Country Hospital - Urology Clinic, Sibiu
  - Oncomed SRL, Timișoara
- Russia (19):
  - Arkhangelsk Regional Oncology Center, Arkhangelsk
  - Chelyabinsk Regional Oncology Center, Chelyabinsk
  - Republican Clinical Oncology Center, Kazan'
  - Kazan City Oncology Center, Kazan'
  - Research Institute of Urology, Moscow
  - Russian Oncological Research Center n.a. N.N. Blokhin, Moscow
  - Russian Research Center of Radiology, Moscow
  - Medical Radiology Research Center, Obninsk
  - Orenburg Regional Clinical Oncology Center, Orenburg
  - Leningrad Regional Oncological Center, Saint Petersburg
  - Municipal Aleksandrovskaya Hospital, Saint Petersburg
  - Municipal Multi-Speciality Hospital #2, Saint Petersburg
  - Municipal Hospital #26, Saint Petersburg
  - Municipal Clinical Oncology Center, Saint Petersburg
  - Central Research Institute of Roentgenology and Radiology, Saint Petersburg
  - Research Institute of Oncology n.a. Professor N.N. Petrov, Saint Petersburg
  - Municipal Hospital #15, Saint Petersburg
  - Stavropol Territorial Clinical Oncology Center, Stavropol
  - Regional Clinical Oncology Hospital, Yaroslavl
- Ukraine (11):
  - Cherkassy Regional Oncology Center, Cherkassy
  - Chernigov Regional Oncology Center, Chernihiv
  - Urology Department, Dnepropetrovsk State Medical Academy, Dnipro
  - City General Hospital #4, Dnipro
  - Donetsk Regional Antitumor Center, Donetsk
  - Ivano-Frankovsk Regional Oncology Center, Ivano-Frankivsk
  - Kharkiv Regional Urology and Nephrology Center, Kharkiv
  - Institute of Urology under the Academy of Medical Sciences of Ukraine, Department of Plastic and Supportive Urology, Kiev
  - Institute of Urology under the Academy of Medical Sciences of Ukraine, Urology Department, Kiev
  - State Regional Diagnostics and Treatment Oncology Center, Lviv
  - Regional Oncology Center, Uzhhorod
- United Kingdom (7):
  - Addenbrooke's Hospital, Cambridge Clinical Trials Centre, Cambridge
  - Derby Hospital NHS Trust, Derby
  - The Beatson West of Scotland Cancer Centre, Glasgow
  - St. James's Institute of Oncology, Leeds
  - The Royal Marsden NHS Trust, London
  - The Christie Hospital NHS Trust, Manchester
  - South Wales Cancer Institute, Singleton Hospital, Swansea

REFERENCES:
- [Result] Hawkins R, Gore M, Shparyk Y, Bondar V, Gladkov O, Ganev T, Harza M, Polenkov S, Bondarenko I, Karlov P, Karyakin O, Khasanov R, Hedlund G, Forsberg G, Nordle Ö, Eisen T. A randomized phase 2/3 study of naptumomab estafenatox plus IFN-α vs IFN-α in advanced renal cell carcinoma. ASCO Annual Meeting 2013; Abstract ID: 3073.
- [Result] Eisen T, Hedlund G, Forsberg G, Nordle Ö, Hawkins R. Baseline biomarker trend analysis of a randomized phase 2/3 study of naptumomab estafenatox plus IFN-α vs IFN-α in advanced renal cell carcinoma. European Cancer Congress (ECCO) 2013; Abstract ID: 2710.
- [Result] Elkord E, Burt DJ, Sundstedt A, Nordle O, Hedlund G, Hawkins RE. Immunological response and overall survival in a subset of advanced renal cell carcinoma patients from a randomized phase 2/3 study of naptumomab estafenatox plus IFN-alpha versus IFN-alpha. Oncotarget. 2015 Feb 28;6(6):4428-39. doi: 10.18632/oncotarget.2922. PMID 25669986
- [Derived] Aldin A, Besiroglu B, Adams A, Monsef I, Piechotta V, Tomlinson E, Hornbach C, Dressen N, Goldkuhle M, Maisch P, Dahm P, Heidenreich A, Skoetz N. First-line therapy for adults with advanced renal cell carcinoma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 May 4;5(5):CD013798. doi: 10.1002/14651858.CD013798.pub2. PMID 37146227